CLINICAL TRIAL: NCT05090982
Title: Creation of a Shared Medical Decision-making Tool for Atopic Dermatitis
Acronym: SHADOW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211198; 2021-A01859-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-09-22; First posted 2021-10-25 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; shared medical decision-making tool; e-Delphi
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Atopic dermatitis: 150 patients with Atopic dermatitis
  Interventions: Other: Audio recordings during the consultations; Other: Audio recordings during the consultations and test of the shared medical decision-making tool for modification; Other: Audio recordings during the consultations and test of the shared medical decision-making tool for validation

INTERVENTIONS:
Other: Audio recordings during the consultations — 50 patients with audio recordings of the consultation
Other: Audio recordings during the consultations and test of the shared medical decision-making tool for modification — 50 patients with audio recording of the consultation and Test of the shared medical decision-making tool for modification
Other: Audio recordings during the consultations and test of the shared medical decision-making tool for validation — 50 patients with audio recording of the consultation and test of the shared medical decision-making tool for validation.

SUMMARY:
Hypothesis/Objective : Patient-centered health care and shared decision making are key components of increasing importance which are recommended by the French Haute Autorite de Sante (HAS) and World Health Organization (WHO).

In the context of dermatology and atopic dermatitis, European guidelines has promoted an active involvement from both patients and caregivers in therapeutic decisions at all stages to achieve therapeutic success and the Task Force on Atopic Dermatitis (ETFAD) has promoted the setting of treatment goals in a shared decision with the patient.

The main objective of this study is to develop and cross culturally validate a tool dedicated to shared-decision in atopic dermatitis that can be used during routine dermatological consultations.

The second objective is to better characterize patients seen in this context and to evaluate patients' satisfaction when empowered by shared decision.

Method : We aim to develop a SDMt in AD following the recommendations of the International Patient Decision Aid Standards (IPDAS) collaboration. Development will use a multistep approach: 1) identification of priority domains for patients; 2) Selection of domains to be included in the SDMt for AD; and 3) Creation and testing of the SDMt.

Participants will be consecutive adult (>18 years old) patients attending consultation for a AD in medical centres in France (Toulouse, Nantes and Créteil). All participants will provide written consent to participate. The study will be submitted for approbation to the local ethics committees of the University Hospital Centres of Paris and will be conducted according to the Declaration of Helsinki.

Step 1: Identification of priority domains for patients

Step 2: Selection of domains to be included in the SDMt for AD

Step 3: Creation and testing of the SDMt

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* Patient with atopic dermatitis
* Written information given to the patient and no objection from the patient to participate to the study

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient with cognitive dysfunction that makes it impossible to communicate effectively or to complete the questionnaire
* Patient under AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Atopic Dermatitis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Creation of a shared medical decision-making tool in the context of a consultation for atopic dermatitis in a specialized dermatology consultation. | through study completion, an average of 1 year
  Qualitative descriptions of the topics discussed by the patient during the therapeutic decision in a specialized dermatology consultation for atopic dermatitis; in other words, to characterize the topics discussed by the patient during the consultation

SECONDARY OUTCOMES:
Patient satisfaction with the therapeutic decision-making process | during the intervention
  SURE satisfaction score
Assessment of the perceived state of the patient about the intervention | during the intervention
  Validation tool score CollaboRATE
Assessment of the psychological state of the patient | during the intervention
  Validation tool score GAD-7
Assessment of the perceived health state of the patient | during the intervention
  Score of PHQ-9 questionnaire
Assessment of the quality of life of the patient | during the intervention
  Score of DLQI questionnaire
Assessment of the stigmatization perceived by the patient | during the intervention
  6-items Stigmatization scale
Assessment of the severity perceived by the patient | during the intervention
  Atopic Dermatitis Perceived Severity Scale
Description of treatment compliance in patients who received the validated tool | during the intervention
  Compliance with treatment received

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-André Natella, PhD, Study Director — Assistance Publique - Hôpitaux Paris
Locations (1):
- Hospital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
APHP IS DATA'S OWNER, PLEASE CONTACT BOARD